CLINICAL TRIAL: NCT00443144
Title: D3-Growth Hormone Receptor Polymorphism and Total Effect of Recombinant Human Growth Hormone on Growth in Girls With Turner Syndrome
Brief Title: D3-GHR Polymorphism and Turner Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Gerhard Binder, Pediatric Endocrinology, University Hospital Tuebingen
Other Study IDs: TS-TUE-FH1
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Turner Syndrome; Short Stature
Keywords: growth hormone receptor polymorphism; pharmacogenomics; growth promoting therapy
MeSH Terms: conditions — Turner Syndrome; Dwarfism | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: recombinant human growth hormone

SUMMARY:
The protein polymorphism of the growth hormone receptor characterized by the genomic deletion of exon 3 has been linked to the magnitude of the first-year-growth response to growth hormone (GH) in girls with Turner syndrome.

Objective: to study the long-term effect of GH therapy in Turner syndrome in correlation to this GHR polymorphism in a mainly retrospective design (chart-review).

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome defined by a structural aberration or lack of the X chromosome.
* Growth velocity less than 2 cm/year at the time of final analysis (= final height).

Exclusion Criteria:

* Age <3.5 or >14 years at start of GH therapy,
* GH peak serum levels < 8 ng/ml in two independent tests,
* Thelarche at start or during the first year of treatment,
* Oxandrolone therapy for any time and a duration of GH therapy less than 2 years.

Ages: 38 Months to 14 Years | Sex: Female
Age Groups: Child
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Binder, M.D. PhD, Principal Investigator — University-Children's Hospital Tübingen
Locations (1):
- University-Children's Hospital, Tübingen, Germany

REFERENCES:
- [Background] Dos Santos C, Essioux L, Teinturier C, Tauber M, Goffin V, Bougneres P. A common polymorphism of the growth hormone receptor is associated with increased responsiveness to growth hormone. Nat Genet. 2004 Jul;36(7):720-4. doi: 10.1038/ng1379. Epub 2004 Jun 20. PMID 15208626